CLINICAL TRIAL: NCT00861510
Title: A Pilot Study of the Safety and Efficacy of Escalating Doses of ON 01910.Na in Patients With Relapsed Mantle Cell Lymphoma, Multiple Myeloma, Chronic Lymphocytic Leukemia, and Related Lymphoid Malignancies
Brief Title: A Pilot Study of the Safety and Activity of Escalating Doses of ON 01910.Na in Patients With Relapsed Mantle Cell Lymphoma, Multiple Myeloma, Chronic Lymphocytic Leukemia, and Related Lymphoid Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 090094; 09-H-0094
Record Dates: First submitted 2009-03-12; First posted 2009-03-13 (Estimated); Last update posted 2019-12-03 (Actual); Status verified 2014-09-04

CONDITIONS: Lymphoma, Mantle-cell; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Hairy Cell; Waldenstrom Macroglobulinemia; Multiple Myeloma
Keywords: Small Lymphocytic Lymphoma (SLL); Prolymphocytic Lymphoma (PLL); Hairy Cell Leukemia (HCL); Mantle Cell Lymphoma; MCL; Chronic Lymphocytic Leukemia; CLL; Multiple Myeloma; MM
MeSH Terms: conditions — Lymphoma, Mantle-Cell; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Hairy Cell; Waldenstrom Macroglobulinemia; Multiple Myeloma | interventions — ON 01910

INTERVENTIONS:
Drug: ON01910 Na

SUMMARY:
Background:

* Mantle cell lymphoma (MCL), chronic lymphocytic leukemia (CLL), multiple myeloma (MM), and other lymphoid malignancies are all incurable lymphoid malignancies that mainly affect persons in their late 60s and early 70s. Conventional chemotherapy can achieve high rates of clinical response, but relapse following these responses is almost universal. Patients with lymphoid malignancies relapse because their tumor cells become resistant to chemotherapy; therefore, new types of drugs are needed for better treatment responses.
* The investigational drug ON 01910.Na has been shown to be active against MCL and CLL cells, but further research is needed to determine the most safe and effective dose for this drug.

Objectives:

* To determine the maximum tolerated dose (the highest dose that does not cause unacceptable side effects) of ON 01910.Na in patients with cancers of the lymphoid cells.
* To study the effects that ON 01910.Na has on cancers of the lymphoid cells.

Eligibility:

* Patients 18 years of age and older who have been diagnosed with cancer of the lymphoid cells, and who have not been able to take or have not benefitted from existing treatment options.

Design:

* Evaluations before the treatment period:
* Full medical history and physical examination, and pregnancy test for women.
* Blood and urine tests.
* Disease evaluation with computerized tomography (CT) scan, magnetic resonance imaging (MRI), electrocardiogram; bone marrow and lymph node biopsies; and skeletal x-rays, if clinically indicated.
* Treatment with ON 01910.Na:
* Different research subjects will receive increasing doses of ON 01910.Na to determine which dose is considered safe.
* To reduce the risk of one rare serious side effect of treatment for myeloid malignancies, patients will take allopurinol 12 hours before and 7 days after each drug infusion, one 300 mg pill each day.
* Cycles 1 2: Patients will be admitted to the clinical center for 2 days at the beginning of each cycle. Each cycle involves intravenous infusion of ON 01910.Na continuously for a period of 48 hours, followed by 12 days of observation. Researchers will try to maintain the schedule of 2 days of infusion every 14 days, but the interval between doses may be extended if patients experience delayed recovery blood counts.
* Cycles 3 4: Patients who are doing well and choose to continue may receive an additional two cycles (2 days of inpatient infusion followed by 12 days of outpatient observation). At the end of cycle 4, researchers will determine if the disease is responding to therapy. Patients who experience side effects may continue to take ON 01910.Na at a lower dose or may stop receiving the drug.
* Patients who respond well to four cycles of ON 01910.Na may be eligible for additional cycles of ON 01910.Na.
* Patients who need to start another medication to treat their disease will stop taking ON 01910.Na, and the researchers will perform a final study visit 2 weeks after the last dose of ON 01910.Na. After that, participation in the study will be complete.

DETAILED DESCRIPTION:
Mantle cell lymphoma (MCL), chronic lymphocytic leukemia (CLL), multiple myeloma (MM) and the related lymphoid malignancies included in this protocol are all incurable lymphoid malignancies that mainly affect persons in their late 60s and early 70s. Conventional chemotherapy can be effective at achieving high rates of clinical response, but relapse following these responses is almost universal. Response rates in the relapsed setting are inferior due to acquired resistance of the tumor cells, and new therapies with novel mechanisms of action are needed. Our aim in this study is to specifically address the needs of these patients for whom few effective treatments are available.

Patients with lymphoid malignancies relapse due to acquired resistance of tumor cells to chemotherapy agents and innovative targeted therapies which overcome these mechanisms of resistance are needed. One such investigational drug, ON 01910.Na, is a potent and selective inhibitor of the cell cycle and leads to reduction in cyclin D1 expression. In vitro, ON01910.Na shows activity against CLL and MCL cell lines with resultant cellular death. The overexpression of cyclin D1 in these related lymphoid malignancies provides a rationale for its use in selected patients with these conditions.

We therefore propose this non-randomized, pilot, dose-escalating Phase I study of ON 01910.Na in patients with MCL, CLL, MM and related lymphoid malignancies who have relapsed after or are refractory to standard therapy.

The primary objective is to determine the toxicity profile (including the maximum tolerated dose and recommended phase II dose) of ON 01910.Na when administered the first 2 (or amended later to 3) days of a 2-week cycle in escalating doses in patients with MCL, CLL, MM and related lymphoid malignancies.

The first cohort was dosed at 1200mg/m2/day times 2 days. The second cohort was dosed at 1500mg/m2/day for 2 days. Three subjects were enrolled into the third cohort at 1800mg/m2/day times 2 days. One subject completed the 1800mg/m2/ day times 2 days dosing scheme. Two subjects stopped study drug after the first dose due to progressive disease. The 3 subjects who received 1800mg/m2/day times 2 days will compose cohort 3. New safety data from the drug manufacturer lead to Amendment L, which changed the dosing from 48 hours to 72 hours. On November 18, 2010, the IRB approved Amendment L, which changed the dosing for the new cohorts 4 and 5 to 1800mg/day times 3 days, and 2100mg/day times 3 days, respectively.

Secondary objectives include, the biological effects of ON 01910.Na (for example cyclin D1 expression) on cell-cycle pathways of cells obtained from blood, lymph nodes or bone marrow, the toxicity profile of ON 01910.Na with subsequent dosing after 2 cycles of therapy, early indications of biologic activity after 4 cycles of therapy, evaluation of the pharmacokinetics of ON 01910.Na at the RPTD level, and indications of biologic activity during extended access (after 4 cycles (day 56)).

The primary endpoint will be the toxicity profile at each dose level through day 28 (cycle 2 day 14).

Secondary endpoints include the reduction in lymph nodes, quantification of circulating lymphoma cells, assessment of extranodal disease sites, and/or measurement of the malignant monoclonal proteins in the serum or urine after 4 cycles of therapy (day 56).

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Histologically documented or cytologically confirmed diagnosis of Mantle Cell Lymphoma (MCL) and refractory to, or relapsed after, greater than or equal to 1 prior lines of antineoplastic therapy (including an anthracycline or mitoxantrone and rituximab, each in one or more lines).

     OR

     Histologically documented or cytologically confirmed diagnosis of Chronic Lymphocytic Leukemia (CLL), Small Lymphocytic Lymphoma (SLL), or Prolymphocytic Lymphoma (PLL) and refractory to, or relapsed after, greater than or equal to 1 prior lines of antineoplastic therapy (including either a nucleoside analogue or an alkylating agent or a combination thereof. Must have relapsed after, failed or opted not to receive rituximab or alemtuzumab. Not a candidate for or opted not to participate in bone marrow transplantation.

     OR

     Histologically documented or cytologically confirmed diagnosis of Multiple Myeloma (MM) and refractory to, or relapsed after greater than or equal to 2 prior lines of antineoplastic therapy including both bortezomib and an immunomodulatory (IMiD) agent such as lenalidomide or thalidomide.

     OR

     Histologically documented or cytologically confirmed diagnosis of Waldenstrom s macroglobulinemia (WM) or Hairy Cell Leukemia (HCL) and refractory to, or relapsed after greater than or equal to 1 line of antineoplastic therapy.
  2. Measurable disease (defined as two dimensional disease on imaging or quantifiable leukemic disease or monoclonal paraproteins).
  3. Failed to respond to, relapsed following, not eligible for, or opted not to participate in other standard of care treatment options.
  4. Age greater than or equal to 18 and less than or equal to 99.

EXCLUSION CRITERIA:

1. Less than 4 weeks since having received any other treatments directed toward their malignancy (standard or investigational). Steroids permissible up to 2 weeks prior to enrollment.
2. Malignant disease other than MCL, CLL/SLL, PLL, WM, HCL or MM requiring treatment with cytotoxic therapy.
3. Active infection not adequately responding to appropriate therapy.
4. HIV positive patients and taking anti-retroviral therapy.
5. Moribund status or concurrent hepatic, renal, cardiac, neurologic, pulmonary, infectious, or metabolic disease of such severity that it would preclude the patient s ability to tolerate protocol therapy.
6. Symptomatic congestive heart failure, unstable angina pectoris, history of life threatening cardiac arrhythmia, myocardial infarction within 6 months or new conduction abnormalities by EKG. Patients with symptoms of coronary artery disease or EKG abnormalities must be evaluated and cleared by cardiology prior to enrollment.
7. Uncontrolled hypertension (defined as systolic pressure greater than or equal to 160 and/or diastolic pressure greater than or equal to 110).
8. New onset seizures (within 3 months prior to the first dose of ON 01910.Na) or poorly controlled seizures.
9. ECOG performance status 3 or 4.
10. Life expectancy less than 3 months.
11. Absolute neutrophil count (ANC) less than 500.
12. Platelet count less than 25,000 micro/L, unless responsive to platelet transfusion so that count can be maintained greater than 10,000 micro/L.
13. Total bilirubin greater than or equal to 1.5 mg/dL not related to hemolysis or Gilbert s disease, ALT or AST greater than or equal to 2 times ULN.
14. Serum creatinine greater than 1.5 times ULN or a calculated creatinine clearance of less than 40 mL/min/1.73 m(2).
15. Ascites requiring active medical management including paracentesis, or hyponatremia (defined as serum sodium value of less than 134 meq/L).
16. Current pregnancy, unwilling to take oral contraceptives or refrain from pregnancy if of childbearing potential or currently breastfeeding.
17. Male patients with female sexual partners who are unwilling to follow the strict contraception requirements described in this protocol.
18. Major surgery within 3 weeks of ON 01910.Na treatment initiation
19. Psychiatric illness/social situations that would limit the patient s ability to tolerate and/or comply with study requirements.
20. Unable to understand the investigational nature of the study or give informed consent.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2009-03-05; Primary Completion 2012-10-19 (Actual); Study Completion 2012-10-19 (Actual)

PRIMARY OUTCOMES:
Safety of escalating doses ON01910.Na at day 28.

SECONDARY OUTCOMES:
The reduction in lymph nodes, quantification of circulating lymphoma cells, assessment of extranodal disease sites, and/or measurement of the malignant monoclonal proteins in the serum or urine after 4 cycles of therapy (day 56).

CONTACTS AND LOCATIONS:
Overall Officials: Mark J Roschewski, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Park IW, Reddy MV, Reddy EP, Groopman JE. Evaluation of novel cell cycle inhibitors in mantle cell lymphoma. Oncogene. 2007 Aug 16;26(38):5635-42. doi: 10.1038/sj.onc.1210350. Epub 2007 Mar 19. PMID 17369860
- [Background] Paul JT, Henson ES, Mai S, Mushinski FJ, Cheang M, Gibson SB, Johnston JB. Cyclin D expression in chronic lymphocytic leukemia. Leuk Lymphoma. 2005 Sep;46(9):1275-85. doi: 10.1080/10428190500158797. PMID 16109604
- [Background] Gumireddy K, Reddy MV, Cosenza SC, Boominathan R, Baker SJ, Papathi N, Jiang J, Holland J, Reddy EP. ON01910, a non-ATP-competitive small molecule inhibitor of Plk1, is a potent anticancer agent. Cancer Cell. 2005 Mar;7(3):275-86. doi: 10.1016/j.ccr.2005.02.009. PMID 15766665